CLINICAL TRIAL: NCT05731921
Title: Investigation of the Effect of the Exercise Program With the 'Empathy Dress' Applied to Midwifery Students on the Levels of Physical Discomfort, Empathy and Compassionate Love: A Randomized Controlled Study
Brief Title: Effect of 'Empathy Dress' and Exercise on Midwifery Students' Discomfort, Empathy and Compassionate Love Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Emine Akca, Assist. Prof. Dr. in the Amasya University Midwifery Department, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Amasya Univ
Record Dates: First submitted 2023-02-09; First posted 2023-02-16 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Empathy; Discomfort; Love
Keywords: Midwifery; Student; Empathy level; Physical discomfort level; Compassionate Love level

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with pretest-posttest control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The exercise program with the 'Empathy Dress'
  Interventions: Behavioral: The exercise program with the 'Empathy Dress'
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: The exercise program with the 'Empathy Dress' — The experimental group will be given an exercise program that includes a total of eight sessions (two months) of 'Empathy Dress' and some exercises (stairs going up and down, sitting up, putting on trousers, tying shoes, etc.), every week and 20 minutes per week, by the researchers.
  Arms: Experimental group

SUMMARY:
To investigate the effect of the exercise program with the 'Empathy Dress' applied to midwifery students on the Levels of physical discomfort, empathy and compassionate love in the midwifery department of Amasya University. A total of 62 midwifery student are planned to be included in the study. Data will be collected with the "Student Information Form", "The Toronto Empathy Questionnaire- TEQ", "Evaluation Scale for Physical Discomfort", and "The Compassionate Love Scale". In the study, an exercise program that includes a total of eight sessions of 'Empathy Dress' and some exercises, every week and 20 minutes per week to the midwifery students in the experimental group, by the researcher. It is thought that the results of the study will improve the empathy and sensitive love levels of midwifery students and increase the quality of midwifery care offered.

DETAILED DESCRIPTION:
Midwifery education consists of two parts, theoretical and clinical, which complement each other. Educators in the field of midwifery should strengthen students' skills before going to the clinic by following innovative training techniques. In this context, it is recommended that the simulation supported midwifery education model be used, disseminated and included in the curriculum of midwifery departments, as it contributes to students.To investigate the effect of the exercise program with the 'Empathy Dress' applied to midwifery students on the Levels of physical discomfort, empathy and compassionate love in the midwifery department of Amasya University. A total of 62 midwifery student (31 experimental, 31 control) are planned to be included in the study. Data will be collected with the "Student Information Form", "The Toronto Empathy Questionnaire- TEQ", "Evaluation Scale for Physical Discomfort", and "The Compassionate Love Scale". In the study, an exercise program that includes a total of eight sessions (two months) of 'Empathy Dress' and some exercises (stairs going up and down, sitting up, putting on trousers, tying shoes, etc.), every week and 20 minutes per week to the midwifery students in the experimental group, by the researcher. The expected result of the study is to determine whether the exercise program with the 'Empathy Dress' is an effective intervention in increasing the empathy and compassionate love levels in midwifery students. In addition, the effect of the 'Empathy Dress' and exercise program on the physical discomfort levels of midwifery students is investigated. It is thought that the results of the study will improve the empathy and sensitive love levels of midwifery students and increase the quality of midwifery care offered.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Absence of a defined psychiatric disorder
* There is no problem that prevents communication

Exclusion Criteria:

* Those who have movement system problems that prevent them from exercising with increasing weights by adapting to their pregnancy weeks,
* Individuals who do not meet the inclusion criteria or who do not volunteer to participate in the research despite meeting them will be excluded from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Midwifery Students
Enrollment: 57 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Empathy Level | 2 months
  Empathy is one of the primary outcomes. This will be measured using 'The Toronto Empathy Questionnaire- TEQ'. The minimum score that can be obtained from the scale is "13", the maximum score is "65", and as the score obtained from the scale increases, empathy levels also increase.
Compassionate Love Level | 2 months
  Compassionate Love Level is the other primary outcomes. This will be measured using 'The Compassionate Love Scale'. The minimum score that can be obtained from the scale is "21", the maximum score is "147", and as the score obtained from the scale increases, Compassionate Love levels also increase.

SECONDARY OUTCOMES:
Physical Discomfort Level | 2 months
  Physical Discomfort Level is the other primary outcomes. This will be measured using 'Evaluation Scale for Physical Discomfort'. This form was developed by the researchers and consists of 4 items. The score ranges from 0 to 10 points, with increasing score reflecting more discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İbici Akça, Ph.D, Principal Investigator — Amasya University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No